CLINICAL TRIAL: NCT07249008
Title: Effects of a Non-sugar Sweetener Label on Parents' Selection of Foods and Beverages in Brazil: a Randomized Clinical Trial.
Brief Title: NSS Grocery Store Brazil
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Responsible Party: Principal Investigator, Allison Sylvetsky (Meni), Associate Professor, Vice Chair of the Department of Exercise and Nutrition Sciences, George Washington University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: FWA00005945
Record Dates: First submitted 2025-09-15; First posted 2025-11-25 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Control Group; Mexico-based NSS FOPL; Brazil-based NSS FOPL

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Participants view the online store without any non-sugar sweetener front-of-package label
- Mexico-based NSS FOPL (Experimental): Participants view the online store with the Mexican-style non-sugar sweetener front-of-package label on eligible products
  Interventions: Other: Experimental : Mexico-based NSS FOPL
- Brazil-based NSS FOPL (Experimental): Participants view the online store with the magnifying glass non-sugar sweetener front-of-package label like the one used in Brazil
  Interventions: Other: Experimental : Brazil-based NSS FOPL

INTERVENTIONS:
Other: Experimental : Mexico-based NSS FOPL — Participants view the online store with the Mexican-style non-sugar sweetener front-of-package label on eligible products
  Arms: Mexico-based NSS FOPL
Other: Experimental : Brazil-based NSS FOPL — Participants view the online store with the magnifying glass non-sugar sweetener front-of-package label like the one used in Brazil
  Arms: Brazil-based NSS FOPL

SUMMARY:
The purpose of this study is to assess the impact of non-sugar sweeteners (NSS) front-of-package labels (FOPL) on Brazilian parents' food and beverage selections for their children. The study includes three arms: 1. no NSS FOPL control group, 2. a group exposed to a NSS FOPL modeled after the Mexican warning label for NSS, and 3. a group exposed to a NSS FOPL using the magnifying glass symbol currently implemented in Brazil for nutrients of public health concern. Participants will be instructed to select products for their child, including one yogurt, three beverages (for breakfast, lunch, and dinner), one granola, and one cereal bar.

ELIGIBILITY:
Eligible participants include:

* Adults aged 20 years or older,
* Living in Brazil
* Parents or guardians of children between 2 and 12 years old
* Primarily responsible for the household grocery shopping (more than 50%)
* Can read and understand Portuguese

Recruitment will occur nationwide through an online panel, with quotas for education, race, and geographic distribution to approximate the national profile.

Individuals will be excluded if

* Not a parent or guardian of a child aged 2-12 years
* Younger than 20 years
* Not primarily responsible for more than half of the household grocery shopping
* Unable to read or understand Portuguese
* Do not provide informed consent.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1068 (Estimated)
Dates: Start 2025-12-08 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of products selected that are unsweetened or low in added sugars | Day 1
  Selection of products that do not contain NSS or added sugars, or that contain added sugars below the FOPL threshold (i.e., less than 10 g per 100 g) for granola and cereal bars.

SECONDARY OUTCOMES:
Percentage of products selected that contain NSS and high added sugars | Day 1
  Selection of products containing both NSS and are high in added sugars, defined as those displaying the FOPL for added sugars (i.e., more than 7.5 g per 100 ml for liquids, and more than 10 g per 100 g for foods).

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-11-19): https://cdn.clinicaltrials.gov/large-docs/08/NCT07249008/Prot_SAP_000.pdf